CLINICAL TRIAL: NCT04295395
Title: Evaluation of the Brain and Renal Regional Oxygenation Using Near Infrared Spectroscopy (NIRS) Method in Very Low Birth Weight (<1500 g) Infants
Brief Title: Evaluation of the Brain and Renal Regional Oxygenation Using NIRS in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Vilnius University (Other)
Responsible Party: Sponsor
Other Study IDs: AIRS-2017
Record Dates: First submitted 2020-02-19; First posted 2020-03-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2021-03

CONDITIONS: Pre-Term; Persistent Ductus Arteriosus
Keywords: near-infrared spectroscopy; preterm infant; echocardiography
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group1: preterm infant with closed ductus arteriosus, <32 weeks birth weight < 1500g, and > 72 hours of age
  Interventions: Device: NONIN SenSmart model X-100 near- infrared spectrometer
- group2: preterm infant with PDA < 32 weeks, birth weight < 1500g, and > 72 hours of age
  Interventions: Device: NONIN SenSmart model X-100 near- infrared spectrometer
- group3: preterm infant with hemodynamically significant PDA < 32 weeks, birth weight < 1500g, and > 72 hours of age
  Interventions: Device: NONIN SenSmart model X-100 near- infrared spectrometer

INTERVENTIONS:
Device: NONIN SenSmart model X-100 near- infrared spectrometer — for to measure cerebral (cSO2) and renal (rSO2 ) regional tissue oxygen saturation on the day after echocardiography was done. The sensors were placed on the right/left forehead and the right/left lateral posterior flank
  Other Names: GE LOGIQ S8 XDclear 2.0 ultrasoud

SUMMARY:
This study evaluates the brain and renal oxygenation using near infrared spectroscopy in preterm infants with persistent ductus arteriosus

DETAILED DESCRIPTION:
Patent ductus arteriosus (PDA) is common in preterm infants. In the presence of a large PDA, significant systemic to pulmonary shunting occurs, which may result in pulmonary hyperperfusion and systemic hypoperfusion.

The evidence on PDA effect on brain and renal tissue oxygenation, measured by Near Infrared Spectroscopy is still controversial.

This study aims to evaluate the brain and renal oxygenation using near infrared spectroscopy (NONIN SenSmart model X-100) in 3 groups of preterm infants: 1) closed ductus arteriosus, 2) persistent ductus arteriosus, 3) hemodynamicaly significant ductus arteriosus.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with gestation age of < 32 weeks
* birth weight < 1500g
* > 72 hours of age.

Exclusion Criteria:

* cardiovascular, renal, cerebral congenital defects,
* confirmed sepsis,
* no parental consent

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants with gestation age of < 32 weeks, birth weight < 1500g, > 72 hours of age, will have NIRS monitors placed to measure cerebral and renal regional tissue oxygenation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Differences of the mean values of regional oxygenation of the brain and renal | from Day 4 of live up to 36 weeks
  Cerebral and renal regional tissue oxygen saturation monitoring on the day after echocardiography was done

CONTACTS AND LOCATIONS:
Overall Officials: Augustina Jankauskiene, MD, Study Director — Vilnius University
Locations (1):
- Vilnius University Santaros Klinikos Neonatology Center, Vilnius, Lithuania

REFERENCES:
- [Derived] Navikiene J, Virsilas E, Vankeviciene R, Liubsys A, Jankauskiene A. Brain and renal oxygenation measured by NIRS related to patent ductus arteriosus in preterm infants: a prospective observational study. BMC Pediatr. 2021 Dec 9;21(1):559. doi: 10.1186/s12887-021-03036-w. PMID 34886825